CLINICAL TRIAL: NCT05816720
Title: Retrospective Analysis of Patients Re-treated With Lutetium-177 DOTATATE (Lutathera®)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA601A1US08
Record Dates: First submitted 2023-01-30; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Initial treatment: Patients who received initial treatment with lutetium-177 DOTATATE
  Interventions: Drug: Lutetium-177 DOTATATE
- Re-treatment: Patients who received re-treatment with lutetium-177 DOTATATE
  Interventions: Drug: Lutetium-177 DOTATATE
- Additional re-treatment: Patients who received additional re-treatment with lutetium-177 DOTATATE
  Interventions: Drug: Lutetium-177 DOTATATE

INTERVENTIONS:
Drug: Lutetium-177 DOTATATE — Intravenous administration
  Other Names: Lutathera®

SUMMARY:
This was a retrospective non-interventional study evaluating the medical records of patients with neuroendocrine tumor (NET) re-treated with lutetium-177 DOTATATE at a single United States institution - the Excel Diagnostics & Nuclear Oncology Center in Houston, Texas. Initial treatment was defined as the initial regimen of up to 4 doses of Lutetium-177 DOTATATE received by each patient; re-treatment was defined as any additional dose(s) of lutetium-177 DOTATATE given after the patient progressed following the initial treatment, with a minimum time interval of 6 months between the initial treatment and re-treatment.

The study period was from 01 January 2010 to 30 June 2021. The index date was the date of the first ever treatment with lutetium-177 DOTATATE, and the index re-treatment date was the date of the first re-treatment dose of lutetium-177 DOTATATE received. The index (identification) period was from 01 July 2010 to 31 December 2020 to account for minimum 6-month baseline and follow-up periods. Patients were followed from the index date to the occurrence of one of the following events (whichever came first):

1. Date of death - the date at which a patient was reported in the database as having died
2. Last month active - the last recorded mention of the patient in the dataset
3. End of data window - end of the dataset Patient characteristics were assessed at both the index date and the index re-treatment date. Real-world effectiveness and safety outcomes were also assessed from the index date and from the index re-treatment date.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of any NET
* Evidence of re-treatment with lutetium-177 DOTATATE

  * Documentation of initial treatment with a regimen of up to 4 doses of lutetium-177 DOTATATE, followed by evidence of progression, and then ≥1 subsequent dose of lutetium-177 DOTATATE
  * Minimum of 6 months between the end of the initial treatment doses and the first re-treatment dose

Exclusion criteria

• <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 11 years
  Time from the index date of treatment or re-treatment with lutetium-177 DOTATATE until the date of progression or death
Overall survival | Up to approximately 11 years
  Time from the index date of treatment or re-treatment with lutetium-177 DOTATATE until the date of death
Percentage of patients with treatment response | Up to approximately 11 years
  Best overall response was defined per Response Evaluation Criteria In Solid Tumors (RECIST), 1.1. Overall response: complete response (CR) + partial response (PR); CR; PR; stable disease (SD); and progressive disease (PD)

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) | Up to approximately 11 years
Mean change from baseline in white blood cell (WBC) count | Up to approximately 11 years
Mean change from baseline in hemoglobin | Up to approximately 11 years
Mean change from baseline in absolute neutrophil count (ANC) | Up to approximately 11 years
Mean change from baseline in lymphocyte count | Up to approximately 11 years
Mean change from baseline in platelet count | Up to approximately 11 years
Mean change from baseline in alkaline phosphatase (ALP) | Up to approximately 11 years
Mean change from baseline in alanine aminotransferase (ALT) | Up to approximately 11 years
Mean change from baseline in aspartate aminotransferase (AST) | Up to approximately 11 years
Mean change from baseline in albumin | Up to approximately 11 years
Mean change from baseline in bilirubin | Up to approximately 11 years
Mean change from baseline in creatinine | Up to approximately 11 years
Mean change from baseline in estimated glomerular filtration rate (eGFR) | Up to approximately 11 years
Mean change from baseline in cromogranin A | Up to approximately 11 years
Mean change from baseline in pancreatic polypeptide | Up to approximately 11 years
Mean change from baseline in pancreastatin | Up to approximately 11 years
Number of patients who received other treatments prior to initial treatment with lutetium-177 DOTATATE | Prior to initial treatment with lutetium-177 DOTATATE
Number of patients who received lutetium-177 DOTATATE, categorized by number of doses | Up to approximately 11 years
Number of patients who received lutetium-177 DOTATATE, categorized by treatment stage | Up to approximately 11 years
Quantity of lutetium-177 DOTATATE administered, categorized by treatment stage | Up to approximately 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Excel Diagnostics & Nuclear Oncology Center, Houston, Texas, United States